CLINICAL TRIAL: NCT02354196
Title: Big PICTURE 2: Physicians International CT Utilization Registry 2
Brief Title: Physicians International CT Utilization Registry 2
Acronym: Big PICTURE 2
Status: Withdrawn | Type: Observational
Sponsor: MDDX LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Big PICTURE 2
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2015-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CCTA: Subjects who underwent a CCTA
  Interventions: Procedure: CCTA

INTERVENTIONS:
Procedure: CCTA — CT of heart to assess coronary disease
  Other Names: Cardiac CT Angiography

SUMMARY:
To determine the total plaque burden, plaque severity and composition of patients undergoing Cardiac CT who do not have any previous history of CVD. There are two cohorts:

1. A retrospective follow-up for MACE endpoints of patients who underwent a CCTA >1 year ago as part of the Big PICTURE Trial, who meet the inclusion criteria of Big PICTURE 2.
2. A prospective observational registry of patients referred to undergo CCTA with a 1 and 2 year follow-up.

DETAILED DESCRIPTION:
In the original BIG PICTURE trial, the analysis of over 6000 subject's CCTA images found significant differences amongst patients of Arabic and south-east Asian descent, with regard to plaque burden, severity and composition. Due to the "all-comers" nature of that trial, the factors of diabetes, previous CVD, and other coronary risk factors were likely confounders in the results. In this trial, those subject selection is screened to eliminate those factors with the goal of working with a more homogenous population to perform the plaque analysis. This study is a multicenter, prospective, post marketing, observational registry study designed to describe frequency and patterns of various risk factors, indications and findings in patients who undergo CCTA.

BIG PICTURE 2 (abbreviated as "BP2") will collect data on patients from a wide variety of imaging sites (inpatient, outpatient, in-clinic CT machine). While the majority of the sites are within the US, the data collection will not be limited to US-only sites. A sub study of BP2 will perform a remote short follow-up questionnaire of subjects who were in the original Big PICTURE study.

ELIGIBILITY:
Subject Inclusion Criteria

* 18 years or older
* No prior CVD
* No hypertension
* No Diabetes
* Body mass index (BMI) <35 kg/m2.

Subject Exclusion Criteria

* <18 years or older
* Prior CVD
* Hypertension
* Body mass index (BMI) >=30 kg/m2.
* Diabetes Mellitus Type 1 or 2
* Current or previous history of smoking
* Pregnancy
* Planned intervention or bypass surgery
* Known complex congenital heart disease
* Planned invasive angiography for reasons other than CAD
* Non-cardiac illness with life expectancy < 2 years
* Inability to provide written informed consent
* Concomitant participation in another clinical trial in which subject is subject to investigational drug or device
* Pregnant women
* Allergy to iodinated contrast agent
* Serum creatinine >1.5 mg/dl or GFR <30 ml/min
* Baseline irregular heart rhythm
* Heart rate ≥100 beats per minute
* Systolic blood pressure ≤90 mm Hg
* Contraindications to β blockers or nitroglycerin Strategies for Recruitment and Retention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1000 subjects, 18 or older, no previous CAD
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Plaque characteristics | Immediately after scan
  Total plaque burden, composition, location, severity and myocardial perfusion deficits

SECONDARY OUTCOMES:
MACE endpoints | 2 years (or more)
  Standard MACE endpoints

CONTACTS AND LOCATIONS:
Locations (2):
- MDDX, San Francisco, California, United States
- FACTS, Hyderabad, India